CLINICAL TRIAL: NCT00816452
Title: Title: Increase Awareness to Osteopenia/Osteoporosis Treatment of Patients With Prostate Cancer, by Bisphosphonate Therapy - Registry.
Brief Title: Awareness to Osteopenia's Treatment by Bisphosphonate in Male Suffering From Prostate Cancer
Acronym: InoPro
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Other Study IDs: RISED_L_04261
Record Dates: First submitted 2008-12-31; First posted 2009-01-01 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Osteoporosis; Prostate Cancer
Keywords: Osteoporosis; Prostate Cancer; Osteoporosis in male with Prostate Cancer
MeSH Terms: conditions — Osteoporosis; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Patients with prostate cancer treated in outpatient clinics will be recruited by their urologist physician.

Primary Objective: To evaluate the compliance in male patients with prostate cancer treated with Bisphosphonate and that suffered from Osteopenia/osteoporosis.

Secondary objectives:

To evaluate the compliance of family physicians to prescribe Bisphosphonate for patients upon recommendation by Urologists.

To evaluate the overall number of patients treated by Bisphosphonate in the out-patient clinics, To evaluate incidence of osteopenia/osteoporosis in this study population.

ELIGIBILITY:
Inclusion Criteria:

* Man with Prostate Cancer
* Men ≥70 years old or ≥60 years old treated by LH-RH agonist for at least 2 years or Man who was diagnosed in the past with Osteopenia/osteoporosis
* Osteopenia/osteoporosis proven by bone density test.

Exclusion Criteria:

* Creatinine clearance < 30ml/min
* Hypercalcemia
* Actual treatment by Bisphosphonate or steroids
* Hypersensibility to Bisphosphonate or any contraindication to its use.
* Metastatic prostate Cancer
* Patients not suitable for compliance.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male with Prostate Cancer suffering from Osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To evaluate the compliance in male patients with prostate cancer treated with Bisphosphonate and that suffered from Osteopenia/osteoporosis. | 6 months

SECONDARY OUTCOMES:
To evaluate the compliance of family physicians to prescribe Bisphosphonate for patients upon recommendation by Urologists. | 6 months
To evaluate the overall number of patients treated by Bisphosphonate in the out-patient clinics | 6 months
To evaluate incidence of osteopenia/osteoporosis in this study population. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nurit Tweezer, Study Director — Sanofi-aventis administrative office Israel
Locations (1):
- Sanofi-aventis administrative office, Netanya, Israel